CLINICAL TRIAL: NCT03968172
Title: Development and Evaluation of a Web-based Lifestyle Intervention for EmPOWERment in Early Multiple Sclerosis (POWER@MS1) - a Randomized Controlled Trial and Mixed-methods Process Evaluation
Brief Title: Interactive Web Platform for EmPOWERment in Early Multiple Sclerosis
Acronym: POWER@MS1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Charite University, Berlin, Germany (Other); University of Cologne (Other); University Medical Center Goettingen (Other); Heinrich-Heine University, Duesseldorf (Other); Gaia AG (Industry); BKK Dachverband e.V. (Unknown); Deutsche Multiple Sklerose Gesellschaft (DMSG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: POWER@MS1
Record Dates: First submitted 2019-05-15; First posted 2019-05-30 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Complex Intervention; Lifestyle Intervention; Randomized Controlled Trial; Evidence-based Medicine
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study will be conducted as an investigator blinded trial and participating physicians as well as MS centres in general will not be provided with any information about the group assignment. Randomisation will take place only after baseline documentation. Blinding of the trial participants is pursued, but only possible to a limited extent. Furthermore, it cannot be prevented that patients discuss the intervention contents with their physician. Thus, participants and neurologist might realize their participation in the intervention group. While blinding in behavioural interventions is virtually not possible, the only strategy to increase similarity of groups is to have an active control group which we aim for with the optimized standard care group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EBBC programme (Experimental): Participants in the intervention group will receive access to evidence-based patient information (EBPI) about lifestyle factors in MS combined with a complex behaviour change programme (EBBC programme), an online tool that was developed in line with principles of patient empowerment and cognitive behavioural therapy (CBT) approaches, including acceptance and mindfulness oriented techniques.
  Interventions: Behavioral: EBBC programme
- Control group programme (Active Comparator): Participants randomized to the active control group will receive access to an information platform with optimized standard care consisting of information compiled from the German Multiple Sclerosis Society (DMSG) information material to reflect current practice.
  Interventions: Behavioral: Control group programme

INTERVENTIONS:
Behavioral: EBBC programme — Web-based behavioural lifestyle intervention that provides patients with coordinated information based on their existing health beliefs, interests, etc. In the programme, techniques and exercises will be taught in sequentially active interactive learning units ("simulated dialogues") and followed-up with email and SMS reminders in the second study year. The following topics will be focused on:
  1. Diagnosis and disease progression
  2. Support in disease processing
  3. Techniques for coping with stress and depressive symptoms as well as developing positive emotions
  4. Optimisation of dietary behaviour
  5. Optimisation of physical activity behaviour
  6. Sleep hygiene and methods for dealing with insomnia.
  The programme will accompany each patient with information material and e-mail reminders over a period of 12 months with initial 2-3 weekly tasks, later only weekly reminders and inputs every 2 weeks. All in all, the intervention programme will consist of 16 modules.
  Arms: EBBC programme
Behavioral: Control group programme — Web-based information platform with optimized standard care compiled from information material of the German Multiple Sclerosis Society (DMSG). Information will be provided in sequentially activated modules over a period of 12 months, covering the following topics:
  1. Disease progression
  2. Invisible symptoms of multiple sclerosis
  3. Symptomatic therapy
  4. Immunotherapy decision support
  5. Coping strategies
  6. Autonomy
  7. Fatigue
  8. Quality of life
  9. Physical activity
  10. Nutritional behaviour
  In addition, a reminder system with neutral e-mail reminders will be used to promote the use of the programme.
  Arms: Control group programme

SUMMARY:
This randomized controlled trial with an accompanying process evaluation investigates the hypothesis that behavioural and web-based information on immunotherapy decisions, disease management and lifestyle can change patient behaviour resulting in reduced inflammatory disease activity in multiple sclerosis.

DETAILED DESCRIPTION:
After a multiple sclerosis (MS) diagnosis, uncertainty and psychological stress may have a negative effect on the disease course, while psychological counselling may reduce inflammatory activity. Therefore, especially newly diagnosed patients require intensive and individual support to deal with the disease and to initiate lifestyle changes. This is hardly available in standard care. Systematic, evidence-based patient information on the value of lifestyle change is not available either.

POWER@MS1 aims to encourage patients with MS to find the best way of dealing with the disease on the basis of evidence-based patient information (EBPI) and a complex behaviour change intervention. The platform will serve as a disease accompanying empowerment programme. Various modules will be provided to accompany patients with MS (pwMS) at an early stage of the disease. The multicomponent intervention will offer comprehensive support after diagnosis, which includes, firstly, an immunotherapy decision-support programme aligned with principles of shared decision-making (SDM), and, secondly, a behaviour-change intervention promoting disease management and lifestyle habits over a period of one year. Ideally, POWER@MS1 leads to a more targeted immunotherapy start, and consequently to better adherence and optimization of a preventive effective lifestyle.

Primary objective:

To determine if a web-based behavioural intervention on immunotherapy decision making, disease management, and lifestyle can reduce the inflammatory disease activity in MS (a relapse or - as a surrogate for inflammatory disease activity - new T2 lesions on magnetic resonance imaging (MRI)).

Secondary objectives:

The secondary objectives are to determine if the web-based intervention can

* strengthen patient autonomy and empowerment,
* promote informed decisions on immunotherapy,
* improve quality of life,
* reduce anxiety and depression,
* increase physical activity and a healthy diet,
* increase effectiveness of neurologists encounters,
* and save health care costs.

In order to develop and evaluate the intervention, a multiphase mixed-methods study covering the first three phases of the Medical Research Council Framework for complex interventions will be conducted. After development, the intervention programme will be pretested and piloted with experts and persons with MS (pwMS). The intervention will be evaluated in a randomized controlled trial (RCT) with 328 patients with early MS (< 12 months), who have at least two MS-typical lesions. Study participants will be recruited in 19 MS centres across Germany and randomised to an intervention group with access to an evidence-based information platform or to a control group with optimised standard care based on material of the German Multiple Sclerosis Society (DMSG). The primary endpoint will be reached if new T2 lesions or relapses occur. Furthermore, a mixed methods process evaluation and a health economic evaluation will be carried out.

Recalculated sample size: Based on a blinded data export of August 16th, 2021, with data on event rates (primary endpoint: new T2 lesion or new relapse) of 135 included patients at that time, a blinded sample size recalculation was performed. The sample size recalculation resulted in a lower number of necessary cases due to high event rates (51 primary endpoint events at that time). The calculation of event rates and an assumed dropout rate of 20% resulted in a case number of 216 patients that have to be randomized (108 per group) instead of 328.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* clinically isolated syndrome (CIS), suspected or confirmed MS for less than 12 months
* at least two MS-typical lesions on T2-weighted images on MRI scans
* MS typical cerebrospinal fluid (CSF) finding with detection of oligoclonal bands
* access to the internet and ability to use websites

Exclusion Criteria:

* corticosteroid therapy within 4 weeks prior to study inclusion
* substantial psychiatric disorder (based on clinical impression)
* severe cognitive deficit affecting information uptake (based on clinical impression)
* pregnancy
* claustrophobia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-04-05 (Actual); Study Completion 2023-04-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of new lesions on T2-weighted images on MRI scans | Change in the number of lesions on T2-weighted images from immediately after patient inclusion (month 0), to month 3, 6, 12, 18 (follow-up) and 24 (follow-up) after patient inclusion
  As a surrogate for inflammatory disease activity, new T2 lesions will be assessed in MRI.
  MRI protocol: Localizer, 3D FLAIR sagittal e.g. 3x3mmm, 3D image T1w native sagittal, 1-3mm, PD/T2w axial 3mm, protocol duration approx. 20 min.
Time to a second relapse | Change in relapse status from baseline (no endpoint), to month 1, 3, 6, 12, 18 (follow-up), and 24 (follow-up) after patient inclusion
  Duration of complaints/impairment, relapse symptoms (worsened or newly occurred), degree of impairment due to the relapse and degree of certainty with regard to the classification of the worsening as a relapse.

SECONDARY OUTCOMES:
Risk Knowledge (RiKno10) | Month 3 after patient inclusion
  To assess risk knowledge, RiKno 2.0 was adapted to a 10-item version (RiKno10).
Control Preference Scale (CPS) | Month 12 after patient inclusion, as well as after reaching the primary endpoint
  As a surrogate of decision quality, preferred and realized role preference based on the Control Preference Scale (CPS) will be assessed. The scores for preferred and realized roles are grouped into active, collaborative or passive.
Immunotherapy Decision Satisfaction Questionnaire | After reaching the primary endpoint
  As a surrogate of decision quality, satisfaction with the immunotherapy decision will be assessed.
Immunotherapy Status Questionnaire | Baseline (no endpoint), month 1, 3, 6, 12, 18 (follow-up), 24 (follow-up) after patient inclusion
  It will be assessed whether an immunotherapy was newly started, aborted or changed.
Patient Activation Measure (PAM) | Baseline and month 12 after patient inclusion
  Assessment of patient activation development (i.e. expressed in the confidence and knowledge to take action, as well as actually taking health-related action).
Coping self-efficacy (CSE) scale | Baseline and month 12 after patient inclusion
  Based on the coping self-efficacy (CSE) scale, selected and adapted items will be used to measure perceived self-efficacy for emotion-focused coping behaviours. In this study, response options are ranging from 0 (completely disagree), representing a low coping self-efficacy value, to 3 (fully agree), representing a high coping self-efficacy value.
Changes in Perceived Empowerment Questionnaire | Month 12 after patient inclusion
  Changes in perceived empowerment will be measured based on selected and adapted items of a 3-point scale empowerment questionnaire measuring changes in patients' feelings of empowerment and/or control over their health problem.
Credibility/Expectancy Questionnaire | 4 weeks after patient inclusion (month 1)
  Selected items measuring treatment expectancy and credibility.
Readiness to Change (stage assessment) based on the Health Action Process Approach (HAPA) | Baseline, month 3 and 12 after patient inclusion
  Readiness to change will be assessed based on the Health Action Process Approach (HAPA) in order to determine the interventions impact on willingness to change lifestyle activities, such as physical activity and nutritional behaviour.
Impairment in the Expanded Disability Status Scale (EDSS) | Baseline and month 12 after patient inclusion
  MS impairment measurement with a score ranging from 0.0 (normal neurological exam) to 10.0 (death due to MS).
Hamburg Quality of life in MS Scale (HAQUAMS) | Baseline and month 12 after patient inclusion
  Assessment of MS-specific quality of life based on 8 subscales (consisting of 38 individual items) and 4 additional questions. For all subscales, averaged subscores are calculated from the values of the respective items (ranging from 1 to 5), with high scores standing for low quality of life and low scores standing for high quality of life.
EQ-5D | Baseline, month 6, 12, 18 (follow-up) and 24 (follow-up) after patient inclusion
  Assessment of health-related quality of life.
Hospital anxiety and distress scale (HADS) | Baseline and month 12 after patient inclusion
  Assessment of depression and anxiety based on 14 items on 2 scales (7 on the subscale "anxiety" and 7 on the subscale "depression"), ranging from 0 (low anxiety/depression level) to 3 (high anxiety/depression level) per item, resulting in a range of 0 to 21 per scale or 0 to 42 for the total HADS value.
Godin Leisure-Time Exercise Questionnaire (GLTEQ) | Baseline and month 12 after patient inclusion
  Amount of mild, moderate and strenuous exercise in leisure time.
Physical Activity, Exercise, and Sport Questionnaire (Bewegungs- und Sportaktivität Fragebogen (BSA-F)) | Baseline and month 12 after patient inclusion
  Assessment of physical activity, including occupational activity, leisure time activity and sports.
Questionnaire of Healthy Diet (QHOD2), adapted version of the Mediterranean Diet Screener (aMDS) | Baseline, month 3 and 12 after patient inclusion
  Frequency of intake of characteristic food groups (e.g. vegetables, fish, and olive oil) in the last seven days and is an indicator of the degree of adherence to an adapted Mediterranean dietary pattern.
24-h dietary recall myfood24 | Baseline and month 12 after patient inclusion, in each case three times within two to three weeks (two weekdays and one weekend day)
  Aggregated nutrient intake data (e.g. omega-3-fatty acids).
Health Economic Evaluation | Baseline, month 6, 12, 18 (follow-up) and 24 (follow-up) after patient inclusion
  Assessment of all direct costs associated with the intervention as well as costs resulting from the consumption of health-related goods and services as well as indirect costs due to productivity losses.

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Heesen, Prof., Principal Investigator — Universitätsklinikum Hamburg-Eppendorf
Locations (1):
- Universitätsklinikum Hamburg-Eppendorf, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
An anonymized individual data set will be published in major journals in order to disseminate the study results. In addition, all trial results will be communicated at scientific conferences and meetings by the investigators and presented on the DMSG website and other relevant patient websites.

REFERENCES:
- [Derived] Krause N, Riemann-Lorenz K, Steffen T, Rahn AC, Pottgen J, Stellmann JP, Kopke S, Friede T, Icks A, Vomhof M, Temmes H, van de Loo M, Gold SM, Heesen C. Study protocol for a randomised controlled trial of a web-based behavioural lifestyle programme for emPOWERment in early Multiple Sclerosis (POWER@MS1). BMJ Open. 2021 Feb 16;11(2):e041720. doi: 10.1136/bmjopen-2020-041720. PMID 33593774

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-07-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT03968172/SAP_000.pdf